CLINICAL TRIAL: NCT02209948
Title: Clinical Trial Phase IIB Randomized, Multicenter, of Continuation or Non Continuation With 6 Cycles of Temozolomide After the First 6 Cycles of Standard First-line Treatment in Patients With Glioblastoma.
Brief Title: Temozolomide 12 Cycles Versus 6 Cycles of Standard First-line Treatment in Patients With Glioblastoma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Investigación en Neurooncología (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEINO 14-01; 2014-000838-39 (EudraCT Number)
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Temozolomide (Experimental): Those patients will take 6 additional Temozolomide cycles
  Interventions: Drug: Temozolomide
- Without treatment (No Intervention)

INTERVENTIONS:
Drug: Temozolomide
  Arms: Temozolomide

SUMMARY:
The purpose of this study is to show if prolonging treatment with temozolomide to 12 cycles improve progression-free survival in patients with glioblastoma included in this study, randomized according to o6-methylguanine-DNA-methyltransferase (MGMT) methylation status and residual disease or not, to receive an additional 6 cycles of temozolomide.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and sign the informed consent document .
2. Age greater than or equal 18.
3. Patients with glioblastoma according to WHO classification (glioblastoma ) who received chemo- radiotherapy and temozolomide -based chemotherapy ( Stupp scheme ) and have completed 6 cycles of adjuvant temozolomide (with or without bevacizumab) in the context of standard treatment without presenting progression of disease.
4. Availability of tumor tissue from the first surgery for centralized histological review , for determining the MGMT study if you have not done in the center of origin. (If they were made in the center of origin the result of the center will be accepted ).
5. Stable dose of dexamethasone in the inclusion never above corticoids dose received in cycle 6 of the adjuvant .
6. Index greater than or equal 60 % Karnofsky.
7. All patients must show no progression of disease in a brain nuclear magnetic resonance (NMR) as defined in RANO established criteria before randomization .
8. Basal NMR study on a maximum of 6 weeks prior to inclusion, in which no progress is observed and is permitted to manage the care 6th cycle ( NMR performed after the 6th cycle of adjuvant is also acceptable as long as no progression was observed).
9. Adequate bone marrow reserve : hematocrit greater or equal 29% , white blood cell> 3,000 , RAN greater or equal 1,500 cells / ul , platelets greater or equal 100,000 cells / ul.
10. Creatinine <1.5 times the upper limit of normal (ULN) of the laboratory performing the analysis.
11. Serum bilirubin <1.5 / ULN; SGOT , SGPT < 2.5 times the upper limit of normal of the laboratory performing the analysis. Serum < 3/ULN alkaline phosphatases .
12. Effective contraceptive method in patients and their partners.

Exclusion Criteria:

1. Less than 5 years of any previous invasive neoplasia. In situ cervical carcinoma or basal cell skin carcinoma accepted.
2. Concomitant treatment with other investigational agents (other concomitant bevacizumab) .
3. Presence of any clinically significant gastrointestinal abnormalities that may affect the decision , transit or absorption of study drug , such as the inability to take medication in tablets by mouth.
4. Presence of any psychiatric or cognitive disorder that limits understanding or written informed consent and / or impair compliance with the requirements of this protocol.
5. Concurrent disease that prevents the continuation of temozolomide treatment.
6. Presence of leptomeningeal dissemination.
7. Pregnant or breastfeeding.
8. Positive patients receiving combination antiretroviral therapy in HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-08-22 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Balañá, M.D., Study Chair — Hospital Germans Trias i Pujol - ICO Badalona; Mª Ángeles Vaz, M.D., Study Chair — Hospital Universitario Ramon y Cajal
Locations (20):
- Spain (20):
  - Hospital Universitari Germans Trias i Pujol/ICO Badalona, Badalona, Barcelona
  - Institut Català d'Oncologia L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Son Espases, Palma de Mallorca, Mallorca
  - Hospital Universitario Sant Joan de Reus, Reus, Tarragona
  - Consorcio Hospitalario Provincial de Castellón, Castellon, Valencia
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital Dr. Josep Trueta de Girona, Girona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Balana C, Vaz MA, Manuel Sepulveda J, Mesia C, Del Barco S, Pineda E, Munoz-Langa J, Estival A, de Las Penas R, Fuster J, Girones R, Navarro LM, Gil-Gil M, Alonso M, Herrero A, Peralta S, Olier C, Perez-Segura P, Covela M, Martinez-Garcia M, Berrocal A, Gallego O, Luque R, Perez-Martin FJ, Esteve A, Munne N, Domenech M, Villa S, Sanz C, Carrato C. A phase II randomized, multicenter, open-label trial of continuing adjuvant temozolomide beyond 6 cycles in patients with glioblastoma (GEINO 14-01). Neuro Oncol. 2020 Dec 18;22(12):1851-1861. doi: 10.1093/neuonc/noaa107. PMID 32328662

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 patients do not meet inclusion criteria. Only 159 patients were randomized
Groups:
- Temozolomide: Temozolomide dose 150/200 mg/m2/d for 5 days every 28 days for 6 cycles (total 12 cycles of adjuvant temozolomide).
- Without Treatment: No treatment (total 6 cycles of adjuvant Temozolomide).
Period: Overall Study
Arm/Group | Temozolomide | Without Treatment
Started | 80 | 79
Recieved Alocated Intervention | 80 | 79
Lost to Follow up | 0 | 1
Discontinued Due to Progression | 31 | 39
Completed (Used for analysis) | 80 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Temozolomide | Without Treatment | Total
Number analyzed (Participants) | 80 | 79 | 159
Age, Continuous [Mean (Inter-Quartile Range); unit: Years] | 60.7 [31 to 79] | 60.4 [29 to 83] | 60.4 [29 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 76
  Male | 42 | 41 | 83
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 80 | 79 | 159
Residual disease (>10mm) [Count of Participants; unit: Participants] — The presence of residual disease (visible on MRI and with at least one lesion bigger than 10mm) at the time of inclusion.
  Participants
    Yes | 41 | 42 | 83
    No | 39 | 37 | 76
Karnofski Performance Status (KPS) index [Count of Participants; unit: Participants] — KPS measures the ability of cancer patients to perform routine tasks. Scores on the KPS range from 0% to 100%. A higher score means that the patient is better able to perform daily activities.
  Participants
    <70% | 2 | 2 | 4
    >=70% | 78 | 77 | 155
Residual Neurological symptom [Count of Participants; unit: Participants]
  Yes | 19 | 8 | 27
  No | 60 | 71 | 131
  NA | 1 | 0 | 1
Dexamethasone (DXM) dose at inclusion [Count of Participants; unit: Participants]
  0 mg | 67 | 70 | 137
  0.5-2 mg | 9 | 6 | 15
  >2 mg | 4 | 3 | 7
Barthel index [Count of Participants; unit: Participants] — Barthel index measures functional independence and residual disability in activities of daily living. Values range from 0 to 5, with lower values indicating more disability.
  Participants
    0 | 12 | 9 | 21
    1 | 68 | 70 | 138
Mini-mental status examinaion (MMSE) [Count of Participants; unit: Participants] — The test evaluates attention, language, memory, orientation, visuospatial proficiency.
  The Mini-mental state examination is scored on a scale of 0-30 with scores > 27 interpreted as normal cognitive status. The lower values are associated to worse cognitive status.
  Participants
    <27 | 16 | 10 | 26
    ≥27 | 51 | 60 | 111
    NP/ND | 13 | 9 | 22
Anticonvulsant therapy [Count of Participants; unit: Participants]
  Yes | 37 | 38 | 75
  No | 43 | 41 | 84
Initial surgery- Treatment at diagnosis. [Count of Participants; unit: Participants]
  Biopsy | 7 | 10 | 17
  Complete resection by post-op MRI) | 28 | 35 | 63
  Complete resection without post-op MRI | 20 | 14 | 34
  Subtotal resection | 25 | 20 | 45
O6-methylguanine DNA methyltransferase (MGMT) Methylation status [Count of Participants; unit: Participants]
  Methylated | 49 | 48 | 97
  Unmethylated | 31 | 31 | 62
Isocitrate dehydrogenase 1 (IDH1) Mutation status [Count of Participants; unit: Participants]
  IDH1-R132 mutated by ICH | 1 | 7 | 8
  IDH1-R132 non mutated by ICH | 71 | 66 | 137
  not determined | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival at 6 Month
Description: Percentage of patients without progression of disease and time between start of treatment and progression of disease.
  The progression disease is defined as the time from the date of randomization to the date of progression defined according to the RANO criteria.
Time Frame: 6 month
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Temozolomide | Without Treatment
Number analyzed (Participants) | 80 | 79
percentage of patients | 61.3 [51.5 to 72.9] | 55.7 [45.8 to 67.8]

2. Secondary Outcome: Number of Participants With Adverse Effects
Description: Total number of patients presenting adverse events, stratified by type of event and grade. Adverse Events of special interest: Only relevant differences in toxicity by arm.
Time Frame: Through the whole study. 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Temozolomide | Without Treatment
Number analyzed (Participants) | 80 | 79
Participants
  Lymphopenia: Grade 1-2 | 52 | 33
  Lymphopenia: Grade 3-4 | 3 | 0
  Lymphopenia: not affected | 25 | 46
  Thrombocytopenia: Grade 1-2 | 36 | 17
  Thrombocytopenia: Grade 3-4 | 2 | 0
  Thrombocytopenia: not affected | 42 | 62
  Nausea and vomiting: Grade 1-2 | 30 | 10
  Nausea and vomiting: Grade 3-4 | 0 | 0
  Nausea and vomiting: not affected | 50 | 69
  Fatigue: Grade 1-2 | 35 | 21
  Fatigue: Grade 3-4 | 0 | 0
  Fatigue: not affected | 45 | 58
  Leucopenia: Grade 1-2 | 29 | 20
  Leucopenia: Grade 3-4 | 1 | 0
  Leucopenia: not affected | 50 | 59

3. Secondary Outcome: Progresion Free Survival Median Values
Description: It will be measured following Response assessment in neuro-oncology (RANO) guidelines: progression-free survival
Time Frame: Through the whole study. 4 years. The median follow up for each patient was 33.4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide | Without Treatment
Number analyzed (Participants) | 80 | 79
months | 9.5 [5.93 to 13.07] | 7.77 [5.70 to 9.83]
Statistical Analysis 1: Comparison: Temozolomide vs Without Treatment; Test type: Other — Log Rank (Mantel-Cox); p = 0.943, Log Rank — Threshold P-value of 0.05

4. Secondary Outcome: Overall Survival
Description: Time between start of treatment and death
Time Frame: Through the whole study. 4 years. The median follow up for each patient was 33.4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide | Without Treatment
Number analyzed (Participants) | 80 | 79
months | 18.2 [16.7 to 23.8] | 23.3 [17.9 to 28.7]
Statistical Analysis 1: Comparison: Temozolomide vs Without Treatment; Test type: Other; p = 0.16, Regression, Cox — Threshold of significance P-value 0.05; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.90 to 1.88]

5. Secondary Outcome: Median Progression-free Survival (PFS) by Arm and MGMT Methylation Status
Description: Median Progression Free Survival depending on treatment arm in patients with MGMT methylation
Time Frame: Through the whole study. 4 years. The median follow up for each patient was 33.4 months
Population: Patients with MGMT methylation
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide | Without Treatment
Number analyzed (Participants) | 49 | 48
months | 11.4 [9.2 to 13.6] | 8.5 [6.5 to 10.4]
Statistical Analysis 1: Comparison: Temozolomide vs Without Treatment; Test type: Other; p = 0.99, Regression, Cox — Threshold for significance P-value 0.05; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.65 to 1.5]

6. Secondary Outcome: Median Overall Survival (OS) by Arm and MGMT Methylation Status
Description: Median OS depending on treatment arm in patients with methylated MGMT
Time Frame: Through the whole study. 4 years. The median follow up for each patient was 33.4 months
Population: Patients with MGMT methylation
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide | Without Treatment
Number analyzed (Participants) | 49 | 48
months | 20.7 [14.7 to 26.7] | 27.1 [20.3 to 33.9]
Statistical Analysis 1: Comparison: Temozolomide vs Without Treatment; Test type: Other; p = 0.13, Regression, Cox — threshold for significance 0.05; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.89 to 2.33]

7. Secondary Outcome: Translational Sub-study - Biomarkers: mutS Homolog 6 (MSH6) Immunoreactivity
Description: partial immunoreactivity of MSH6 in patients by treatment arm. Tumor samples were stained by immuno-histochemical techniques.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Temozolomide | Without Treatment
Number analyzed (Participants) | 80 | 79
Participants
  MSH6 partial immunoreactivity | 5 | 6
  no MSH6 partial immunoreactivity | 75 | 73

ADVERSE EVENTS:
Time Frame: Through the clinical study. About 4 years
Description: In addition, clinically relevant changes on physical examination and abnormal parameters found on complementary examinations (eg radiography, ECG) should also be reported like Adverse Event (AE).
Arm/Group | Temozolomide | Without Treatment
All-Cause Mortality (participants affected / at risk) | 63/80 | 52/79
Serious Adverse Events (participants affected / at risk) | 9/80 | 5/79
Other Adverse Events (participants affected / at risk) | 80/80 | 79/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=80) | Without Treatment (N=79)
Dysarthria (Nervous system disorders) | 0 | 1 (1)
Neurological impairment (Nervous system disorders) | 2 (2) | 0
Syncope (General disorders) | 0 | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Intracraneal hypertension (Vascular disorders) | 1 (1) | 0
Epileptic crisis (Nervous system disorders) | 1 (1) | 0
Respiratory infection (Infections and infestations) | 1 (1) | 0
Claudication (Cardiac disorders) | 1 (1) | 0
Femur fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
General deterioration (General disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0
Pulmonary embolism (Vascular disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=80) | Without Treatment (N=79)
Leukopenia (Blood and lymphatic system disorders) | 30 (30) | 20 (20)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 8 (8)
Lymphopenia (Blood and lymphatic system disorders) | 55 (55) | 33 (33)
Thrombocytopenia (Blood and lymphatic system disorders) | 38 (38) | 17 (17)
Creatinine high (Renal and urinary disorders) | 3 (3) | 6 (6)
Alkaline Phosphatase High (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Potasium High (Blood and lymphatic system disorders) | 3 (3) | 6 (6)
Sodium High (Blood and lymphatic system disorders) | 7 (7) | 5 (5)
GGT High (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
GOT High (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
GPT High (Blood and lymphatic system disorders) | 5 (5) | 7 (7)
Bilirubin High (Blood and lymphatic system disorders) | 7 (7) | 8 (8)
Hyperglicemia (Metabolism and nutrition disorders) | 14 (14) | 19 (19)
Neurologic (Nervous system disorders) | 38 (38) | 41 (41)
Nausea and Vomiting (Gastrointestinal disorders) | 30 (30) | 10 (10)
Asthenia (General disorders) | 35 (35) | 21 (21)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Skin disorders (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Anxiety (Nervous system disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 13 (13) | 10 (10)
Constipation (Infections and infestations) | 6 (6) | 2 (2)
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 11 (11) | 5 (5)
Thromboembolism (Vascular disorders) | 0 (0) | 2 (2)
Bone Events (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Cardiac Events (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Our trial was not powered to detect significant differences in PFS or OS. To do so, we would have had to know the survival distribution for patients who complete the standard six cycles without progression, but this information was not available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT02209948/SAP_000.pdf
  • Study Protocol (2014-09-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT02209948/Prot_001.pdf